CLINICAL TRIAL: NCT05731856
Title: Impact of Heart Rate Variability Modulation on Stress and Recovery Among Physicians
Brief Title: Impact of Heart Rate Variability Modulation on Stress Management Among Physicians
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Michelle Thompson (Other)
Collaborators: The Board of Medicine (Other); Apollo Neuroscience, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Michelle Thompson, Faculty in Department of Family Medicine, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: STUDY22060130
Record Dates: First submitted 2023-02-09; First posted 2023-02-16 (Actual); Last update posted 2025-10-15 (Actual); Status verified 2025-10

CONDITIONS: Burnout, Professional
MeSH Terms: conditions — Burnout, Professional

STUDY DESIGN:
Intervention Model Description: This is a single group study. All participants will receive identical instructions regarding the device and will complete the same survey measures.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Apollo Intervention Arm (Experimental): Eligible UPMC Physicians and Residents who consent to be part of this study will use an Apollo Device TVS (10-200 Hz) attached to the subject's wrist or ankle via a commercially available wearable vibration technology that can deliver TVS (Transcutaneous Vibratory Stimulation). The intensity will be targeted for the sensory threshold (the level at which the vibration is just noticeable), as this is where the TVS seems most effective from prior studies. Similar vibratory stimuli have been demonstrated to be safe in the literature. The intensity of the vibration will be adjusted to the subjects' comfort and can be controlled by the subject at any time.
  Interventions: Device: Apollo Wearable

INTERVENTIONS:
Device: Apollo Wearable — Participants will be provided with the Apollo wearable device and asked to install the study mobile application on their mobile phones. Participants will use the Apollo for at least 30 minutes after waking up and at least 30 minutes before bed on the corresponding settings for those times of the day. They will be given the Apollo Device TVS (10-200 Hz) to borrow, which they will be instructed to wear daily. They will be asked to wear the device until all study data is collected.
  Other Names: Apollo Neuro

SUMMARY:
The purpose of this research is to examine a wearable device called Apollo that emits gentle vibrations found to benefit mood, energy, and focus. We want to understand how it affects burnout in physicians.

DETAILED DESCRIPTION:
This study will be conducted by using a Tuned Vibroacoustic Stimulation (TVS) device(the commercially available TVS device known as the Apollo wearable), that has been shown in clinical studies at University of Pittsburgh to improve heart rate variability and recovery under stress. The Apollo wearable generates low volume sound waves that feel like a soothing touch to the skin. This study will assess whether slight modulation of heart rate variability (HRV) will result in a reduction in stress, improved recovery, and recovery in and around the hospital. Physicians will wear the Apollo device for heart rate variability modulation and complete questionnaires before and after use of the Apollo device for comparison of outcomes.

ELIGIBILITY:
Inclusion Criteria:

* UPMC attending physicians and residents. The participants must have either IOS or Android phones.

Exclusion Criteria:

* Unwillingness or inability to participate in the study
* Currently own an Apollo device

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2024-01-15 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Copenhagen Burnout Inventory | Through study completion, on average 8 weeks
  The Copenhagen Burnout Inventory (CBI) is a 19-item self reported measure of burnout. It contains three sub-scales measuring personal burnout, work-related burnout, and client-related burnout
Perceived Stress Scale (PSS-10) | Through study completion, on average 8 weeks
  The Perceived Stress Scale (PSS) is the most widely used psychological instrument for measuring the perception of stress using a 10-item survey.
  It is a measure of the degree to which situations in one's life are appraised as stressful.

SECONDARY OUTCOMES:
The Quick Inventory of Depressive Symptomatology | Through study completion, on average 8 weeks
  The QIDS is a brief, 16-item self-rated assessment tool used to evaluate the symptoms of depression present in a patient during the past week.
Pittsburgh Sleep Quality Index (PSQI) | Through study completion, on average 8 weeks
  The Pittsburgh Sleep Quality Index (PSQI) is a self-rated questionnaire which assesses sleep quality and disturbances over a 1-month time interval. With a range of scores 1-21.

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Thompson, DO, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No